CLINICAL TRIAL: NCT00005966
Title: Phase III Randomized Trial of Interferon-Alfa2b Alone Versus Interferon-Alfa2b Plus Thalidomide in Patients With Previously Untreated Metastatic or Unresectable Renal Cell Carcinoma
Brief Title: Interferon Alfa-2b With or Without Thalidomide in Treating Patients With Metastatic or Unresectable Kidney Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067949; ECOG-2898
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2002-09

CONDITIONS: Kidney Cancer
Keywords: stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Interferon-alpha; Thalidomide

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: thalidomide

SUMMARY:
RATIONALE: Interferon alfa-2b may interfere with the growth of the cancer cells. Thalidomide may stop the growth of cancer by stopping blood flow to the tumor. It is not yet known if interferon alfa-2b is more effective with or without thalidomide in treating kidney cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of interferon alfa-2b with or without thalidomide in treating patients who have previously untreated metastatic or unresectable kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall and progression-free survival at 24 weeks in patients with previously untreated metastatic or unresectable renal cell carcinoma treated with interferon alfa-2b with or without thalidomide.
* Compare the safety of these 2 regimens in these patients.
* Compare the quality of life of patients treated with these 2 regimens.
* Compare the pharmacodynamic effects of these regimens on pharmacodynamic measurements of angiogenesis such as serum and plasma angiogenic factor levels in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to prior nephrectomy (yes vs no), disease-free interval (no more than 1 year vs more than 1 year), and ECOG performance status (0 vs 1 or 2). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive interferon alfa-2b subcutaneously (SC) twice daily beginning on day 1.
* Arm II: Patients receive interferon alfa-2b as in arm I and oral thalidomide once daily beginning on day 1.

Treatment in both arms continues in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response (CR) continue treatment for 24 weeks past CR.

Quality of life is assessed prior to randomization and then every 4 weeks through week 24.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 346 patients (173 per arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven previously untreated metastatic or unresectable renal cell carcinoma

  * Retroperitoneal lymph nodes that are unresectable or those that are not resected at the investigator's discretion are considered metastatic disease
  * Prior nephrectomy allowed provided there is evidence of unresponsive metastatic disease after surgery or within one month prior to study enrollment
* Bidimensionally measurable disease

  * Measurable disease must be outside any prior radiotherapy port
* No history of brain metastases unless surgically resected or treated with gamma knife radiotherapy and currently without radiologic evidence of CNS disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Hemoglobin at least 9 g/dL (transfusion allowed)
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 3 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No myocardial infarction within the past 6 months

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 effective methods of contraception (1 highly active method and 1 barrier method) for at least 4 weeks before, during, and for at least 4 weeks after study participation
* No other malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No uncontrolled diabetes or any other concurrent illnesses that would increase risk
* No history of peripheral neuropathy
* No severe depression

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy (including adjuvant interferon alfa therapy), cellular therapy, or vaccine therapy for renal cell carcinoma
* No prior antiangiogenesis therapy for renal cell carcinoma
* Immunotherapy for prior malignancy allowed (except for interferon alfa therapy)

Chemotherapy:

* No prior chemotherapy for renal cell carcinoma
* Chemotherapy for prior malignancy allowed

Endocrine therapy:

* No prior hormonal therapy for renal cell carcinoma

Radiotherapy:

* See Disease Characteristics
* At least 2 weeks since prior radiotherapy and recovered

Surgery:

* See Disease Characteristics

Other:

* More than 7 days since prior IV antibiotics for infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10; Primary Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Gordon, MD, Study Chair — Virginia G. Piper Cancer Center at Scottsdale Healthcare - Shea
Locations (14):
- United States (11):
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center-Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Midlands Cancer Center at Midlands Community Hospital, Papillion, Nebraska
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Comprehensive Cancer Center at Our Lady of Mercy Medical Center, The Bronx, New York
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
- Westmead Hospital, Westmead, New South Wales, Australia
- Instituto de Enfermedades Neoplasicas, Lima, Peru
- San Juan City Hospital, San Juan, Puerto Rico

REFERENCES:
- [Result] Gordon MS, Manola J, Fairclough D, et al.: Low dose interferon-α2b (IFN) + thalidomide (T) in patients (pts) with previously untreated renal cell cancer (RCC). Improvement in progression-free survival (PFS) but not quality of life (QoL) or overall survival (OS). A phase III study of the Eastern Cooperative Oncology Group (E2898). [Abstract] J Clin Oncol 22 (Suppl 14): A-4516, 386s, 2004.